CLINICAL TRIAL: NCT02604979
Title: The Influences of Long Periods of Pneumoperitoneum and Head up Position on the Variation of Heart-rate Corrected QT Interval During Robotic-assisted Laparoscopic Gastrectomy - Observational Study
Status: Completed | Type: Observational
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Other Study IDs: 4-2015-0607
Record Dates: First submitted 2015-10-01; First posted 2015-11-16 (Estimated); Last update posted 2017-01-25 (Estimated); Status verified 2017-01

CONDITIONS: Stomach Cancer
MeSH Terms: conditions — Stomach Neoplasms

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Sympathetic activity could be increased during robot-assisted laparoscopic gastrectomy, which is performed in a head up position under CO2 pneumoperitoneum.

Stimulation of the sympathetic nervous system prolongs the QT interval and can increases the susceptibility to life threatening cardiac arrhythmias.

Thus the investigators decided to evaluate the heart-rate corrected QT interval (QTc interval) during robotic-assisted laparoscopic gastrectomy.

ELIGIBILITY:
Inclusion Criteria:

1. ASA class I-II
2. obtaining written informed consent from the patients who were undergoing robot- assisted laparoscopic gastrectomy.

Exclusion Criteria:

1. emergency operation
2. cardiac disease (unstable angina, congestive heart failure, valvular heart disease)
3. ventricular conduction abnormality
4. prior pacemaker insertion
5. abnormal electrolyte values
6. patients who take antiarrythmic agent
7. hepatic or renal failure
8. drug hyperactivity
9. neurological or psychiatric illnesses

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who were undergoing robot- assited laparoscopic gastrectomy
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2015-09-23 (Actual); Primary Completion 2016-02-06 (Actual); Study Completion 2016-02-06 (Actual)

PRIMARY OUTCOMES:
Evaluate the heart-rate corrected QT (QTc) interval (msec) during robotic-assisted laparoscopic gastrectomy | through study completion, an average of 5 hours
  (T0: Pre-induction T1: 10min after anesthetic induction T2: 1min after CO2 pneumoperitoneum T3: 5min after CO2 pneumoperitoneum T4: 30min after steep trendelenburg position T5:60min after steep trendelenburg T6: 90min after steep trendelenburg T7: Supine positon following end of pneumoperitoneum T8: 5 min after end of pneumoperitoneum T9: End of surgery T10: 10min after extubation)

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Anesthesiology and Pain Medicine, Yonsei University College of Medicine, Seoul, Seoul, South Korea

REFERENCES:
- [Derived] Kim NY, Bai SJ, Kim HI, Hong JH, Nam HJ, Koh JC, Kim HJ. Effects of long periods of pneumoperitoneum combined with the head-up position on heart rate-corrected QT interval during robotic gastrectomy: an observational study. J Int Med Res. 2018 Nov;46(11):4586-4595. doi: 10.1177/0300060518786914. Epub 2018 Jul 20. PMID 30027782